CLINICAL TRIAL: NCT00595062
Title: Quadrant High Dose Rate Intraoperative Radiation Therapy (IORT) for Early-Stage Breast Cancer: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-101
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer
Keywords: Breast; Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Radiation: Intra Operative Radiation Therapy (IORT)

INTERVENTIONS:
Radiation: Intra Operative Radiation Therapy (IORT) — Quadrant High Dose Rate Intra Operative Radiation Therapy (IORT)

SUMMARY:
This study was started to validate the possibility of administering radiation therapy during surgery to the tissue surrounding the tumor once the tumor has been removed. This surrounding breast tissue is at greater risk for developing breast recurrences. This treatment may be as effective as the conventional 5-6week radiation treatment in reducing the risk of further local recurrences after breast-conserving surgery.

Through this study, we would like to confirm that this procedure is a safe alternative to conventional breast radiation, with no additional side effects when compared with the conventional surgery and radiation therapy.

DETAILED DESCRIPTION:
This pilot trial will evaluate the feasibility of intra operative radiation therapy (IORT) given in one fraction at the time of wide local excision as the only adjuvant radiation treatment in a group of patients with early-stage invasive breast cancer.

This study will enroll 60 women, older than 60 years of age, with breast cancer not more than 2 cm in size and without evident additional tumoral foci around the tumor or in other areas of the breast. An MSK radiologist will review your mammography to be sure you qualify for this study. You may be asked to undergo additional mammography or other examinations, such as breast ultrasound in order to verify that the tumor is located in a single quadrant of the breast. Some of these procedures are routinely performed in all candidates for conservative breast surgery.

ELIGIBILITY:
Inclusion Criteria:

* Core biopsy or prior open biopsy to establish the diagnosis.
* Over age 60.
* No physical or imaging evidence of multicentricity or multifocality.
* Size equal or less than 2.0 cm radiographically, clinically node negative.
* Patients scheduled for breast conserving surgery

Exclusion Criteria:

* Patients younger than 61 years
* Patients with evidence of multicentric or multifocal disease seen on imaging (mammography )
* Patients with a lesion exceeding 2 cm radiographically
* Paget's disease or pure DCIS without invasive ductal carcinoma
* Histotype not inclusive of ductal carcinoma
* Condition precluding radiation therapy
* Condition precluding regular follow-up
* Evident dimpling of the skin above the tumor
* Usual contraindications for BCS

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2002-10; Primary Completion 2006-01 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To determine tissue tolerance of the breast to a single intraoperative course of radiation. | 7 years
To establish feasibility of the technique in the operating room. | 7 years

SECONDARY OUTCOMES:
overall survival | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Beryl McCormick, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org